CLINICAL TRIAL: NCT00290329
Title: Multicentric, Surveillance Study to Monitor Safety of GSK Biologicals' Purified Meningococcal Polysaccharide Vaccine of Serogroups ACWY in 3,000 Filipino Subjects Aged Above 2 Years When Administered According to the Prescribing Information.
Brief Title: Safety of Purified Meningococcal Vaccine With Serogroups ACWY, in 3,000 Filipino Subjects Aged > 2 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 208144/002
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2017-01

CONDITIONS: Infections, Meningococcal
Keywords: Safety; Meningococcal disease; Meningitidis serogroups A, C,W & Y diseases; Meningococcal vaccine
MeSH Terms: conditions — Meningococcal Infections | interventions — PsACWY vaccine

ARMS (1):
- Group A (Experimental)
  Interventions: Biological: Mencevax ACWY

INTERVENTIONS:
Biological: Mencevax ACWY — 1 subcutaneous injection.
  Other Names: Neisseria meningitidis serogroups A; C; W and Y vaccine

SUMMARY:
GlaxoSmithKline Philippines has submitted a registration file for its Purified Meningococcal Polysaccharide of Serogroup ACWY Vaccine (Mencevax ACWY). This study is being conducted to collect clinical data in the local target population in order to assess the occurrence of rare adverse events after vaccination as per the requirement of Philippines Bureau of Food and Drugs Directive.

DETAILED DESCRIPTION:
All subjects will receive a single dose of GSK Biologicals' Mencevax ACWY vaccine according to the prescribing information. Subjects will be stratified into the following age groups:

2 to 5 years 6 to 17 years > 18 years The Protocol Posting has been updated in order to comply with the FDA Amendment Act, September 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parent/guardian can and will comply with the requirements of the protocol.
* A Filipino male or female > 2 years of age at the time of the first vaccination.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Written informed consent obtained from the subject and/or from the parent/ guardian of the subject.

Exclusion criteria:

* Subjects suffering from acute severe febrile illness.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Pregnant or lactating female.
* Female planning to become pregnant.
* History of chronic alcohol consumption and/or intravenous drug abuse.
* Any contraindications as stated on the Prescribing Information.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2006-01-14; Primary Completion 2006-10-01 (Actual); Study Completion 2006-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Philippines (8):
  - GSK Investigational Site, Alabang, Muntinlupa City
  - GSK Investigational Site, Binangonan, Rizal
  - GSK Investigational Site, Cainta, Rizal
  - GSK Investigational Site, City of Muntinlupa
  - GSK Investigational Site, Las Piñas
  - GSK Investigational Site, Los Banos, Laguna
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Pasay

RESULTS

PARTICIPANT FLOW:
Groups:
- Mencevax ACWY 2-5 YOA Group: Filipino male or female subjects, between and including 2 to 5 years of age, received a single dose of the Mencevax ACWY vaccine, administered by subcutaneous injection in the deltoid region of the arm.
- Mencevax ACWY 6-17 YOA Group: Filipino male or female subjects, between and including 6 to 17 years of age, received a single dose of the Mencevax ACWY vaccine, administered by subcutaneous injection in the deltoid region of the arm.
- Mencevax ACWY ≥ 18 YOA Group: Filipino male or female subjects, aged 18 or older, received a single dose of the Mencevax ACWY vaccine, administered by subcutaneous injection in the deltoid region of the arm.
Period: Overall Study
Arm/Group | Mencevax ACWY 2-5 YOA Group | Mencevax ACWY 6-17 YOA Group | Mencevax ACWY ≥ 18 YOA Group
Started | 102 | 86 | 61
Completed | 102 | 86 | 61
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mencevax ACWY 2-5 YOA Group | Mencevax ACWY 6-17 YOA Group | Mencevax ACWY ≥ 18 YOA Group | Total
Number analyzed (Participants) | 102 | 86 | 61 | 249
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.0 (1.11) | 9.6 (2.80) | 32.5 (10.98) | 12.51 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 45 | 46 | 144
  Male | 49 | 41 | 15 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  East/ South-east Asian | 94 | 73 | 56 | 223
  South Asian | 8 | 13 | 5 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Severe (Grade 3) Unsolicited Adverse Events
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Grade 3 AE = an AE which prevented normal, everyday activities.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax ACWY 2-5 YOA Group | Mencevax ACWY 6-17 YOA Group | Mencevax ACWY ≥ 18 YOA Group
Number analyzed (Participants) | 102 | 86 | 61
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Adverse Events
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site (Mencevax ACWY 2-5 YOA Group) and beyond 50 millimeters (mm) of injection site (Mencevax ACWY 6-17 YOA Group and Mencevax ACWY ≥ 18 YOA Group).
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax ACWY 2-5 YOA Group | Mencevax ACWY 6-17 YOA Group | Mencevax ACWY ≥ 18 YOA Group
Number analyzed (Participants) | 102 | 86 | 61
Participants
  Any Pain | 18 | 10 | 9
  Grade 3 Pain | 0 | 0 | 0
  Any Redness | 8 | 0 | 3
  Grade 3 Redness | 0 | 0 | 0
  Any Swelling | 6 | 2 | 0
  Grade 3 Swelling | 0 | 0 | 0

3. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Grade 3 irritability = crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite = not eating at all. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax ACWY 2-5 YOA Group
Number analyzed (Participants) | 102
Participants
  Any Drowsiness | 7
  Grade 3 Drowsiness | 0
  Related Drowsiness | 7
  Any Fever | 3
  Grade 3 Fever | 0
  Related Fever | 3
  Any Irritability | 4
  Grade 3 Irritability | 0
  Related Irritability | 4
  Any Loss of appetite | 2
  Grade 3 Loss of appetite | 0
  Related Loss of appetite | 2

4. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], gastrointestinal symptoms and headache. Any = occurrence of the symptom reported irrespective of intensity grade and causal relationship to vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax ACWY 6-17 YOA Group | Mencevax ACWY ≥ 18 YOA Group
Number analyzed (Participants) | 86 | 61
Participants
  Any Fatigue | 1 | 0
  Grade 3 Fatigue | 0 | 0
  Related Fatigue | 1 | 0
  Any Fever | 1 | 0
  Grade 3 Fever | 0 | 0
  Related Fever | 1 | 0
  Any Gastrointestinal symptoms | 1 | 1
  Grade 3 Gastrointestinal symptoms | 0 | 0
  Related Gastrointestinal symptoms | 1 | 0
  Any Headache | 1 | 3
  Grade 3 Headache | 0 | 0
  Related Headache | 1 | 3

5. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax ACWY 2-5 YOA Group | Mencevax ACWY 6-17 YOA Group | Mencevax ACWY ≥ 18 YOA Group
Number analyzed (Participants) | 102 | 86 | 61
Participants | 14 | 9 | 1

6. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 to Month 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mencevax ACWY 2-5 YOA Group | Mencevax ACWY 6-17 YOA Group | Mencevax ACWY ≥ 18 YOA Group
Number analyzed (Participants) | 102 | 86 | 61
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-vaccination period; Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period; SAEs: during the entire study period (from Day 0 to Month 1).
Arm/Group | Mencevax ACWY 2-5 YOA Group | Mencevax ACWY 6-17 YOA Group | Mencevax ACWY ≥ 18 YOA Group
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/86 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/86 | 0/61
Other Adverse Events (participants affected / at risk) | 24/102 | 10/86 | 11/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mencevax ACWY 2-5 YOA Group (N=102) | Mencevax ACWY 6-17 YOA Group (N=86) | Mencevax ACWY ≥ 18 YOA Group (N=61)
Pain (General disorders) | 18 | 10 | 9
Redness (General disorders) | 8 | 0 | 3
Swelling (General disorders) | 6 | 2 | 0
Drowsiness (General disorders) | 7 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.